CLINICAL TRIAL: NCT06346236
Title: Neurodevelopmental Impact of Treatment in Hypothyroxinaemia of Prematurity.
Acronym: NEO-TYR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0843; 401 (Other: AGORA HCL)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Transient Hypothyroxinemia of Prematurity
Keywords: transient hypothyroxinaemia of prematurity, THOP, preterm, prematurity, neurodevelopment, L-thyroxine, ASQ score
MeSH Terms: conditions — Premature Birth | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- THOP treated: Level of circulating T4 < 12 pmol/L at any time of life associated, on the same date, with a level of circulatingon thyro-stimulating hormone < 15 mUI/L if the sample was realiszed before or on the fifteenth day of life OR < 58 mUI/L if the sample was realiszed after the fifteenth day of life, and L-thyroxine treatment is recorded in the medical record (at any dose and with any duration)
  Interventions: Drug: L-thyroxine at a dose of 7.5 µg/kg/d for THOP
- THOP un-treated: Level of circulating T4 < 12 pmol/L at any time of life associated, on the same date, with a level of circulation thyro-stimulating hormone < 15 mUI/L if sample was realiszed before or on the fifteenth day of life OR < 5 mUI/L if sample was realiszed after the fifteenth day of life, and no L-thyroxine treatment recorded in the medical record.
  Interventions: Other: THOP without treatment
- No-THOP: all level of circulating T4 > 12 pmol/L at any time in life
  Interventions: Other: NoTHOP

INTERVENTIONS:
Drug: L-thyroxine at a dose of 7.5 µg/kg/d for THOP — Subjects diagnosed with THOP (as previously defined) and treated with L-thyroxine at a dose of 7.5 µg/kg/d are less likely to have an impaired ASQ score at 4 years of corrected age.
  Groups: THOP treated
Other: THOP without treatment — Subjects diagnosed with THOP (as previously defined) and who received no L-thyroxine treatment.
  Groups: THOP un-treated
Other: NoTHOP — Subjects diagnosed no-THOP (as previously defined)
  Groups: No-THOP

SUMMARY:
Nowadays, taking care of preterm birth is associated with an important increase in survival. This increased survival comes with impairment in neurodevelopmental outcomes in long term evaluation. Thyroid hormones are essentials for brain development, especially for neuronal differentiation. Transient hypothyroxinaemia of prematurity (THOP) is a frequent condition defined by decreased thyroid hormones without the expected rise in thyroid stimulating hormone. Various studies have showed various results regarding the consequences of THOP on neurodevelopment in premature neonates. However, the biggest and most powerful studies agree to say that THOP impair neurodevelopment. On the other hand, only a few studies evaluated the impact of treatment of THOP, and only two focused on treating exclusively the neonates with a biological diagnosis of THOP (Suzumura and co. in 2010 and Nomura and co. in 2014) and their results are inconsistent.

In this study, we aim to show that a treatment with L-thyroxine at a dose of 7.5 µg/kg/j for neonates diagnosed with THOP (defined as a level of l-T4 < 12 pmol/L and a level of TSH < 15 mUI/L before 15 days of life or < 85 mUI/L after 15 days of birth) is associated with an increased neurodevelopmental prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born before or at 3032 weeks of gestation
* For whom blood sample for thyroid examination has been performed for routine care during his stay in neonatology unit.

Exclusion Criteria:

* Other type of thyroid dysfunction (including, but not exclusively: mother with Basedow disease, congenital hypothyroidism, hyperthyroidism)
* Associated polymalformative sindrome

Max Age: 2 Weeks | Sex: All
Age Groups: Child
Study Population: Reanimation and intensive care units of neonatology in Auvergne-Rhone Alpes region (Lyon Croix Rousse hospital, Lyon Femme mère Enfant hospital, St Etienne Hopital Nord, Grenoble Hopital couple enfant).
Sampling Method: Non-Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Neuro-development judged " abnormal " by the paediatrician during the two years of corrected age's consultation. | Evaluation at two years of corrected age.
  Neuro-development is evaluated routinely by paediatricians during consultation, and this evaluation is reported in medical files.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - HFME, Bron
  - CHU Grenoble, Grenoble
  - CHU Saint EtienneHopital, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided